CLINICAL TRIAL: NCT06108765
Title: Acute Kidney Injury in Poly Trauma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar ibrahim abd elsalam, Emergency medicine residency, Assiut University
Other Study IDs: Acute kidney injury in trauma
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Kidney Injury
Keywords: Polytrauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify the incidence and the factors associated with acute kidney injury in adult poly trauma patients

DETAILED DESCRIPTION:
Trauma causes significant morbidity and mortality in all age groups but particularly for those below 60 years and is one of the top 5 causes of death (1,2).Most deaths occur in adults who are between 15 and 44 years(3).Polytrauma originates from the Greek words poly which means multiple and trauma which means wounds. The term polytrauma, which was defined using the new Berlin definition, as cases with an Abbreviated Injury Scale (AIS)≥3 for two or more different body regions and one or more additional variables from five physiologic parameters (hypotension[systolic blood pressure≤90 mmHg], unconsciousness[Glasgow Coma Scale score≤8], acidosis [base excess≤ -6.0], coagulopathy [partial thromboplastin time≥40 s or international normalized ratio≥1.4], and age [≥70 years]) [4].There are complex pathophysiological changes that happen in a polyrauma patient which requires effective treatment for improving morbidity and mortality outcomes. Hemorrhage, systemic inflammatory response syndrome (SIRS) and multiple organ dysfunction syndrome (MODS) are some of the complications of trauma whose effects are not only local but also systemic. There are mechanisms and triggers which result in cardio-vascular shock, hemostasis, apoptosis, organ dysfunctions and immune suppression (CHAOS) [5]. These local and systemic pathophysiological changes that occur in polytrauma (CHAOS) eventually lead to Acute Kidney Injury (AKI) which further worsens their outcomes [6,7].

ELIGIBILITY:
Inclusion Criteria:

* The present study will be conducted on patients with multiple trauma of both genders "without intently selected certain gender" who have no previous history of kidney disease or chronic illness.

Exclusion Criteria:

* • Patients who are less than 16 years old.

  * Patients with preexisting kidney disease or localized individual trauma.
  * patients with diabetes and hypertension.
  * Patients Post cardiac arrest
  * patients leaving the hospital on the same day or transferred to a different hospital will be excluded from this study.
  * patients refusing study will be excluded.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult polytrauma patients above 16 years old with no history of renal disease or chronic illness
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the incidence of acute kidney injury in poly trauma patients | 7 days
  To identify the incidence and factors associated with acute kidney injury in adult polytrauma patients

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ibrahim, Study Director — Assiut University

REFERENCES:
- [Background] Lopes JA, Jorge S. The RIFLE and AKIN classifications for acute kidney injury: a critical and comprehensive review. Clin Kidney J. 2013 Feb;6(1):8-14. doi: 10.1093/ckj/sfs160. Epub 2012 Jan 1. PMID 27818745